CLINICAL TRIAL: NCT05409040
Title: Health Promoting Lifestyle Behaviors and Associated Factors Among Sohag University Students
Brief Title: Health Promoting Lifestyle Behaviors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rahma Ibrahim Mahmoud, demostrator of public health and community department at Sohag university, Egypt, Sohag University
Other Study IDs: Soh-Med-22-06-03
Record Dates: First submitted 2022-04-10; First posted 2022-06-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthy Life Style

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the Health-promoting Lifestyle behaviors of Sohag University students. Identify socio-demographic determinants of the Health-promoting Lifestyle behaviors

DETAILED DESCRIPTION:
Health is the most fundamental criterion on which man's life is dependent, and it has always been an issue throughout history. Health, according to a definition by the World Health Organization (WHO), is physical, spiritual, mental, social, emotional, and occupational tranquility, and not just the absence of illness. This definition, moreover, has been reintroduced as "people's social and economic potency and dynamicity".

Lifestyle is one of the most important determinants of health promotion that is influenced by cultural, economic, political and religious factors. Lifestyle includes day-to-day behaviors and functions of individuals in job, activities, fun, and diet.

According to WHO, 60% of related factors to individual health and quality of life are correlated to lifestyle .

Millions of people follow an unhealthy lifestyle. Hence, they encounter illness, disability and even death. Problems like metabolic diseases, joint and skeletal problems, cardio-vascular diseases, hypertension, overweight, violence and so on, can be caused by an unhealthy lifestyle. The relationship of lifestyle and health should be highly considered.

Globally, Non-communicable diseases NCDs are the leading cause of premature deaths and chronic disabilities and are responsible for almost 70% of all deaths worldwide.

ELIGIBILITY:
Inclusion Criteria:

Under graduate students in all grades of four randomly selected faculties include 2 practical faculties and 2 theoretical faculties during their academic year 2022/2023 who accept to participate in the study

Exclusion Criteria:

Students who refuse to participate in the study

Ages: 18 Years to 26 Years | Sex: All
Age Groups: Adult
Study Population: under graduate students of Sohag university selected randomly from 4 faculties during their academic year 2022/2023
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Health Promoting Lifestyle Behaviors and associated factors among Sohag University students | 2 months
  Assess the Health-promoting Lifestyle behaviors using Health Promoting Lifestyle Profile II:
  The HPLP II tool consists of 52 health-promoting behavior items that are categorized into six subscales: health responsibility (nine items), spiritual growth (nine items), physical activity (eight items), interpersonal relationships (nine items), nutrition (nine items), and stress management (eight items).
  A Likert-type scale was used to measure each behavior, with ranges of never (1), sometimes (2), frequently (3), and routinely (4).
  The total score of the HPLP II ranges from 52 to 208 and is measured by the mean score of the responses to all 52 HPLP items. The total HPLP II score is further classified into four levels: poor for the range 52-90, moderate for the range 91-129, good for the range 130-168, and excellent for the range 169-208. High scores in every subscale mean more frequent health-promoting behaviors.

SECONDARY OUTCOMES:
Health Promoting Lifestyle Behaviors and associated factors among Sohag University students | 2 months
  Identify socio-demographic determinants of the Health-promoting Lifestyle behaviors using Socio-demographic items (age, gender, marital status, field of study, year of university, place of residence, people live with, number of family member, father education, mother education, father job, mother job, parents' marital status, , economic status ,source of participant's outcome, height, weight, history of chronic disease, history of psychiatric disease, history of psychiatric problem last year, physical activity, perception of health status, number of water cups per day, number of days of eating outside per week, smoking)

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Abd EL-Hameed Ali, Assist professor, Study Director — supervisor